CLINICAL TRIAL: NCT03718845
Title: Evaluation of a Mind-Body Medicine Curriculum for High School Peer Counselors
Brief Title: A Mind-Body Medicine Curriculum for Peer Counselors
Status: Completed | Type: Observational
Sponsor: The Center for Mind-Body Medicine (Other)
Collaborators: Silicon Valley Community Foundation (Other)
Responsible Party: Principal Investigator, James S. Gordon, M.D., Founder and Director, The Center for Mind-Body Medicine
Other Study IDs: BCPS-001
Record Dates: First submitted 2018-10-08; First posted 2018-10-25 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Anxiety
Keywords: Empathy; Hope
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peer Counselors: Mind-Body Medicine Curriculum
  Interventions: Behavioral: Mind-Body Medicine Curriculum

INTERVENTIONS:
Behavioral: Mind-Body Medicine Curriculum — The Mind-Body Medicine curriculum consists of presentations on different mind-body techniques as well as the research supporting the use of these techniques.The mind-body technique is then practiced in a supportive small group setting. Mind-body techniques will include guided imagery, relaxation techniques, several forms of meditation, autogenic training and biofeedback.
  Other Names: Mind-Body Skills Groups

SUMMARY:
This study will evaluate a Mind-Body Medicine curriculum for high school peer counselors in order to answer the following research questions:

1. Will peer counselor participation in the Mind-Body Medicine curriculum increase their sense of self-regulation, responsibility, social competence, and empathy; decrease anxiety; and increase hope?
2. What are the experiences of peer support counselors participating in the Mind-Body Medicine curriculum?

DETAILED DESCRIPTION:
The study will be done at the Marjory Stoneman Douglas High School. The research will use a mixed-methods design by collecting both quantitative and qualitative data. The quantitative data will be in the form of standardized research instruments and the qualitative data will be gathered through focus group interviews with the peer-counselors.

ELIGIBILITY:
Inclusion Criteria:

• All high school students who are participating in the Peer Counseling Program at Marjory Stoneman Douglas High School

Exclusion Criteria:

• None (as long as the students meet the inclusion criteria)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: High school students who are participating in the Peer Counseling Program at Marjory Stoneman Douglas High School
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in State-Trait Anxiety Inventory (STAI) scores | baseline, approximately 2 months, approximately 8 months
  The State-Trait Anxiety Inventory has two subscales: State Anxiety and Trait Anxiety. Each has a minimum score of 20 and a maximum score of 80. Higher scores indicate more anxiety which is a worse outcome.

SECONDARY OUTCOMES:
Change in the Social Emotional Assets and Resilience Scales for Adolescents (SEARS-A) | baseline, approximately 2 months, approximately 8 months
  The Social Emotional Assets and Resilience Scales for Adolescents (SEARS-A) has a total score and four subscales. The score ranges are as follows: Total Score 0-105; Self-Regulation 0-24; Social Competence 0-30; Empathy 0-33; Responsibility 0-18. Lower scores indicate a worse outcome. Subscales are summed to obtain the total score.
Change in the Adult Hope Scale | baseline, approximately 2 months, approximately 8 months
  The Adult Hope Scale has a total score and 2 subscales. The score ranges are as follows: Total Score 8-24; Agency subscale 4-32; Pathways subscale 4-32. Lower scores indicate a worse outcome. Subscales are summed to obtain the total score.

OTHER OUTCOMES:
Focus Group Interviews | baseline, approximately 2 months, approximately 6 months, and approximately 8 months
  Focus group interviews will be held with approximately 3 groups of 8 students to obtain information about the experiences of peer support counselors participating in the Mind-Body Medicine curriculum.

CONTACTS AND LOCATIONS:
Overall Officials: James S Gordon, MD, Principal Investigator — The Center for Mind-Body Medicine
Locations (1):
- Marjory Stoneman Douglas High School, Parkland, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The Center for Mind-Body Medicine website — http://www.cmbm.org